CLINICAL TRIAL: NCT07164638
Title: Lung Ultrasound Versus Inferior Vena Cava Collapsibility Index for Early Prediction of Volume Overload During Transurethral Resection of Prostate: A Prospective Observational Study
Brief Title: Lung Ultrasound Versus Inferior Vena Cava Collapsibility Index for Early Prediction of Volume Overload During Transurethral Resection of Prostate
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shereen Ashraf Abdelrazik El-Sabry, Resident, Tanta University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 36264MS733/11/24
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-11

CONDITIONS: Lung Ultrasound Score; Transurethral Resection (TUR) Syndrome; Prostate
Keywords: Lung Ultrasound; Inferior Vena Cava Collapsibility Index; Overload during Transurethral Resection; Prostate
MeSH Terms: conditions — Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: lung ultrasound (LUS) group (Experimental): Serial lung ultrasound will be performed to patients enrolled in this study before the beginning of the surgery, every 15 minutes in the first 30 minutes, and then every 30 minutes for the rest of the operation.
  Interventions: Procedure: lung ultrasound (LUS)
- Group II: IVC collapsibility index group (Experimental): Serial assessment of IVC collapsibility will be used as a monitoring of volume overload in patients enrolled in this study.
  Interventions: Procedure: IVC collapsibility index

INTERVENTIONS:
Procedure: lung ultrasound (LUS) — Serial lung ultrasound will be performed to patients enrolled in this study before the beginning of the surgery, every 15 minutes in the first 30 minutes, and then every 30 minutes for the rest of the operation.lung ultrasound will be used as a tool for monitoring of EVLW to identify early the subclinical pulmonary edema and ensure timely and correct diagnosis and appropriate management.
  Arms: Group I: lung ultrasound (LUS) group
Procedure: IVC collapsibility index — Serial assessment of IVC collapsibility will be used as a monitoring of volume overload in patients enrolled in this study. Basal IVC scanning using ultrasound will be performed before the start of the operation and serial IVC scanning will be done during the procedure every 15 minutes in the first 30 minutes, and then every 30 minutes for the rest of the operation.
  Arms: Group II: IVC collapsibility index group

SUMMARY:
The aim of this study is to compare between accuracy of lung US and IVC CI for early prediction of volume overload during TURP.

Primary outcome:

The incidence of volume overload during transurethral resection of prostate.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia and its associated symptoms affect many men worldwide, the prevalence is over 210 million men. Up to 50% of men over the age of 50 and up to 80% of men over the age of 80 experience lower urinary tract symptoms from Benign prostatic hyperplasia. Transurethral resection of the prostate is considered the gold standard treatment for prostatic hyperplasia. Small amounts of irrigation fluid are absorbed through the prostatic sinuses in almost every Transurethral resection of the prostate operation. Circulating one liter of irrigation within one hour results in an acute decrease in serum sodium concentration from five to eight mmol/L and may indicate an increased risk of Transurethral resection of the prostate syndrome. Both hypertension and hypotension can be observed in TURP syndrome. Hypertension and reflex bradycardia are explained by rapid volume expansion reaching 200 mL/min. Patients also may develop pulmonary edema due to acute circulatory overload. Transurethral resection of the prostate syndrome is a complication characterized by a change in symptoms from asymptomatic hyponatremia to fatigue, vomiting, confusion, loss of vision, Electrocardiogram changes, seizures, coma, and death. It usually happens due to absorption of irrigation fluid during Transurethral resection of the prostate . This syndrome is related to the amount of fluid entering the circulation through the blood vessels or excessive absorption in the resection area. Increased systolic pressure elevates the left ventricular after load, resulting in heart failure or pulmonary edema, which is characterized by dyspnea, hypoxia, tachypnea and crackles on chest auscultation. Studies have shown that symptomatic heart failure occurs in 1.1% of Transurethral resection of the prostate cases, with severe pulmonary edema occurring in 0.3%. Pulmonary edema is a serious complication of Transurethral resection of the prostate and a common cause of death. The incidence of Transurethral resection of the prostate syndrome is about 3.8% following Transurethral resection of the prostate for Benign prostatic hyperplasia. Most of the studies reports similar incidence of this complication of Transurethral resection of the prostate syndrome in a range of 0-10%. Classic methods for clinical assessment of the patient capacity status, such as central venous pressure monitoring, the Flotrac/Vigileo system, are all invasive and carry risks such as hematoma, pneumothorax, infection, and embolism. In recent years, some non-invasive capacity assessment techniques have been gradually applied, such as lung ultrasound and the inferior vena cava collapsibility index. The aim of this study is to compare between accuracy of lung ultrasound score and inferior vena cava collapsibility index for early prediction of volume overload during TURP.

Primary outcome:

The incidence of volume overload during transurethral resection of prostate.

Secondary outcomes:

The incidence of transurethral resection of prostate.

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* American Society of Anesthesiologists classification II-III
* scheduled for Transurethral resection of the prostate syndrome under spinal anesthesia.

Exclusion Criteria:

* Patient refusal.
* Uncooperative patients.
* Patients with major respiratory, cardiac, renal or hepatic disorders.
* Patients whose ultrasound did not clearly show the inferior vena cava as (morbidly obese patients or patients with moderate to marked ascites).
* Patients who have contraindications to spinal anesthesia (neurological disease, severe hypotension, coagulopathy, low fixed cardiac output).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
incidence of volume overload | 2 HOURS

SECONDARY OUTCOMES:
ABG (PaO2 and O2 saturation) | 2 HOURS

CONTACTS AND LOCATIONS:
Overall Officials: Shereen El-Sabry, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No